CLINICAL TRIAL: NCT07184944
Title: A Multicenter, Multinational, Randomized, Double-blind, Placebo-controlled Phase 3, Maintenance Study to Evaluate the Efficacy and Safety of Duvakitug in Participants With Moderately to Severely Active Crohn's Disease
Brief Title: A Maintenance Study to Investigate the Efficacy and Safety of Duvakitug in Participants With Moderately to Severely Active Crohn's Disease
Acronym: STARSCAPE-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC18327; 2025-521037-86 (Registry Identifier: CTIS); U1111-1314-5471 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Duvakitug dose 1 (Experimental): Subcutaneous (SC) injection as per protocol
  Interventions: Drug: Duvakitug
- Du vakitug dose 2 (Experimental): SC injection as per protocol
  Interventions: Drug: Duvakitug
- Du vakitug dose 3 (Experimental): SC injection as per protocol
  Interventions: Drug: Duvakitug
- Placebo (Placebo Comparator): SC injection as per protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duvakitug — Pharmaceutical form:Injection solution-Route of administration:SC injection
  Other Names: SAR447189
  Arms: Du vakitug dose 2; Du vakitug dose 3; Duvakitug dose 1
Drug: Placebo — Pharmaceutical form:Injection solution-Route of administration:SC injection
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, maintenance, Phase 3 study to evaluate the efficacy and safety of duvakitug in participants with moderately to severely active Crohn's Disease (CD). Study details include:

The study duration may be up to 286 weeks including:

* 40-week Pivotal Maintenance Sub-Study
* 240-week Open-Label Extension (OLE) Sub-Study
* 45-day Follow-Up visit

Note: For the participants who do not enroll into OLE Sub-Study, the duration will be up to 46 weeks, including the 40-week maintenance period and a 45-day follow-up visit.

The treatment duration may be up to 280 weeks including:

* 40 weeks in the Pivotal Maintenance Sub-Study
* 240 weeks in OLE Sub-Study

The total number of on-site visits will be up to 43: - 21 visits in the Pivotal Maintenance Sub-Study - 22 visits in the OLE Sub-Study

ELIGIBILITY:
Inclusion Criteria:

Participants aged ≥18 and ≤80 years of age at Baseline. (Where locally permissible, participants 16 to <18 years of age who meet the definition of Tanner stage 5 for development) Pivotal Maintenance Sub-Study: Participants who achieved clinical response and completed endoscopy at the end of STARSCAPE-1 OLE Sub-Study: Participants who complete the Pivotal Maintenance Sub-Study or participation in the TV48574-IMM-20038 Study

Exclusion Criteria:

Participants with medical or compliance conditions that are deemed unsuitable for the study by the investigator Participants with a known hypersensitivity to duvakitug that makes the participant unsuitable for the study by the investigator The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 671 (Estimated)
Dates: Start 2026-01-29 (Estimated); Primary Completion 2029-08-13 (Estimated); Study Completion 2034-03-20 (Estimated)

PRIMARY OUTCOMES:
Co-primary endpoints US/FDA: Pivotal Maintenance Sub-Study Cohort 1 Proportion of participants achieving clinical remission (CDAI) at Week 40 | Week 40
  Clinical Remission by Crohn's Disease Activity Index (CDAI): CDAI score <150. The CDAI is a measure of disease activity based on symptoms, signs, and a laboratory test. Scores on the CDAI scale range from 0 to 600, with scores below 150 indicating relative disease quiescence (remission), 150 to 219 indicating mild disease activity, 220 to 450 indicating moderate activity, and scores exceeding 450 indicating severe disease.
Proportion of participants achieving Endoscopic Response (SES-CD) at Week 40 | Week 40
  The SES-CD is a standardized method for evaluating disease activity. Score ranges from 0 to 56, where higher scores represent more severe disease. Endoscopic Response by SES-CD is a decrease in SES-CD ≥50% from Baseline (or a decrease of at least 2 points for participants with a Baseline score of 4 or more, and isolated ileal disease) based on central reading.
Co-primary endpoints EU/EMA: Pivotal Maintenance Sub-Study Cohort 1 Proportion of participants achieving clinical remission per PRO-2 at Week 40 | Week 40
  Clinical Remission 2-item patient-reported outcome (PRO-2): average daily stool frequency (SF) ≤3 and not worse than the Baseline, and average daily abdominal pain (AP) ≤1 and not worse than the Baseline.

SECONDARY OUTCOMES:
Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants achieving CDAI clinical response Week 40 | Week 40
  The CDAI is a measure of disease activity based on symptoms, signs, and a laboratory test. Scores on the CDAI scale range from 0 to 600, with scores below 150 indicating relative disease quiescence (remission), 150 to 219 indicating mild disease activity, 220 to 450 indicating moderate activity, and scores exceeding 450 indicating severe disease. Clinical Response by CDAI: decrease in CDAI score of 100 points or more from Baseline.
Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants achieving SES-CD endoscopic remission at Week 40 | Week 40
  The SES-CD is a standardized method for evaluating disease activity. Score ranges from 0 to 56, where higher scores represent more severe disease. Endoscopic remission: a SES-CD ≤4 points (SES-CD ≤2 points for isolated ileal disease) and a SES-CD decrease ≥2 points with no SES-CD sub score >1 point from Baseline.
US/FDA Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants achieving CDAI clinical remission and endoscopic remission at Week 40 | Week 40
  The CDAI is a measure of disease activity based on symptoms, signs, and a laboratory test. Scores on the CDAI scale range from 0 to 600, with scores below 150 indicating relative disease quiescence (remission), 150 to 219 indicating mild disease activity, 220 to 450 indicating moderate activity, and scores exceeding 450 indicating severe disease. The SES-CD is a standardized method for evaluating disease activity. Score ranges from 0 to 56, where higher scores represent more severe disease. Clinical Remission by CDAI: CDAI score <150. Endoscopic remission: a SES-CD ≤4 points (SES-CD ≤2 points for isolated ileal disease) and a SES-CD decrease ≥2 points with no SES-CD sub score >1 point from Baseline.
EU/EMA Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants achieving PRO-2 clinical remission and endoscopic remission at Week 40 | Week 40
  Clinical Remission PRO-2: average daily stool frequency (SF) ≤3 and not worse than the Baseline, and average daily abdominal pain (AP) ≤1 and not worse than the Baseline. The SES-CD is a standardized method for evaluating disease activity. Score ranges from 0 to 56, where higher scores represent more severe disease. Endoscopic remission: a SES-CD ≤4 points (SES-CD ≤2 points for isolated ileal disease) and a SES-CD decrease ≥2 points with no SES-CD sub score >1 point from Baseline.
US/FDA Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants achieving PRO-2 clinical remission at Week 40 | Week 40
  Clinical Remission PRO-2: average daily stool frequency (SF) ≤3 and not worse than the Baseline, and average daily abdominal pain (AP) ≤1 and not worse than the Baseline.
EU/EMA Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants achieving CDAI clinical remission at Week 40 | Week 40
  Clinical Remission by CDAI: CDAI score <150. The CDAI is a measure of disease activity based on symptoms, signs, and a laboratory test. Scores on the CDAI scale range from 0 to 600, with scores below 150 indicating relative disease quiescence (remission), 150 to 219 indicating mild disease activity, 220 to 450 indicating moderate activity, and scores exceeding 450 indicating severe disease.
US/FDA Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants achieving corticosteroids free CDAI clinical remission at Week 40 | Week 40
  Clinical Remission by CDAI: CDAI score <150 and without corticosteroid use for CD for at least 12 weeks prior to assessment. The CDAI is a measure of disease activity based on symptoms, signs, and a laboratory test. Scores on the CDAI scale range from 0 to 600, with scores below 150 indicating relative disease quiescence (remission), 150 to 219 indicating mild disease activity, 220 to 450 indicating moderate activity, and scores exceeding 450 indicating severe disease.
EU/EMA Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants achieving corticosteroids free PRO-2 remission at Week 40 | Week 40
  Clinical Remission PRO-2: average daily stool frequency (SF) ≤3 and not worse than the Baseline, and average daily abdominal pain (AP) ≤1 and not worse than the Baseline and without corticosteroid use for CD for at least 12 weeks prior to assessment.
Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants achieving ulcer-free endoscopy (in the subset of participants with ulcers at Baseline) at Week 40 | Week 40
US/FDA Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants achieving clinical remission per CDAI at Week 40 in the subset of participants with clinical remission per CDAI at Week 0 (maintenance of clinical remission per CDAI) | Week 40
  Clinical Remission by CDAI: CDAI score <150. The CDAI is a measure of disease activity based on symptoms, signs, and a laboratory test. Scores on the CDAI scale range from 0 to 600, with scores below 150 indicating relative disease quiescence (remission), 150 to 219 indicating mild disease activity, 220 to 450 indicating moderate activity, and scores exceeding 450 indicating severe disease.
EU/EMA Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants achieving clinical remission per PRO-2 at Week 40 in the subset of participants with clinical remission per PRO-2 at Week 0 (maintenance of clinical remission per PRO-2) | Week 40
  Clinical Remission PRO-2: average daily stool frequency (SF) ≤3 and not worse than the Baseline, and average daily abdominal pain (AP) ≤1 and not worse than the Baseline.
Pivotal Maintenance Sub-Study Cohort 1: Change from Baseline in PROMIS-Fatigue Short Form 7a T-score at Week 40 | Baseline, Week 40
  The PROMIS Fatigue Short Form 7a uses a 5-point Likert scale for each of its 7 items, resulting in a raw score range of 7 to 35. This raw score is then converted into a T-score, with a mean of 50 and a standard deviation of 10, based on US national norms. Higher T-scores indicate greater fatigue.
Pivotal Maintenance Sub-Study Cohort 1: Change from Baseline in IBDQ total score at Week 40 | Baseline, Week 40
  Inflammatory Bowel Disease Questionnaire (IBDQ) instrument consist of 32 items exploring 4 dimensions: "bowel symptoms" (10 items), "systemic symptoms" (5 items), "emotional function" (12 items) and "social function" (5 items). The total IBDQ total score ranges from 32 to 224 with higher score indicating better quality of life.
Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants with no bowel urgency by NRS at Week 40 | Week 40
  Numeric Rating Scale (NRS) for bowel urgency measures the severity of bowel urgency-the sudden or immediate need to have a bowel movement-experienced in the past 24 hours. This tool utilizes an 11-point scale for evaluation, where 0 represents "no urgency" and 10 signifies the "worst possible urgency".
Pivotal Maintenance Sub-Study Cohort 1: Incidence of CD related hospitalization by Week 40 | Week 0 through Week 40
Pivotal Maintenance Sub-Study Cohort 1: Serum concentrations of duvakitug measured over time | Week 0 through Week 40
Pivotal Maintenance Sub-Study Cohort 1: Incidence of treatment-emergent antidrug antibody (ADA) against duvakitug | Week 0 through Week 40
Pivotal Maintenance Sub-Study Cohort 1: Incidence of treatment-emergent adverse events (TEAEs), TEAE of special interest (TEAESIs), TE serious adverse events (TESAEs) and TEAEs leading to permanent study intervention discontinuation | Week 0 through 45 days after last dose
Open-Label Extension Sub-Study: Incidence of TEAEs, TEAESIs, TESAEs, and TEAEsleading to permanent study intervention discontinuation | Week 40 of pivotal maintenance through 45 days after last dose

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Precision Clinical Research-Site Number: 8400059, Coral Springs, Florida
  - Regis Clinical Research, LLC-Site Number: 8400041, Miami, Florida
  - Correa Research Center-Site Number: 8400010, Miami, Florida

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org